CLINICAL TRIAL: NCT06316024
Title: Early Oral Intake of Different Types of Diets Affecting Gastrointestinal Function During Postpartum Recovery After Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Early Oral Intake of Different Types of Diets Affecting Gastrointestinal Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2023056
Record Dates: First submitted 2024-01-04; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-02

CONDITIONS: Cesarean Section
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nothing Per Os group (No Intervention): The participants do not drink anything approximately 6-8 hours after surgery.
- water group (Experimental): The participants drink 240 ml water approximately 6-8 hours after surgery.
  Interventions: Dietary Supplement: water
- juice/sport drink group (Experimental): The participants drink 240 ml juice/sport drink approximately 6-8 hours after surgery.
  Interventions: Dietary Supplement: juice/sport drink group
- chewing gum group (Experimental): The participants start chewing gum approximately 6-8 hours after surgery.
  Interventions: Dietary Supplement: Chewing gum group

INTERVENTIONS:
Dietary Supplement: water — The participants drink 240 mL of water approximately 6-8 hours after surgery
  Arms: water group
Dietary Supplement: juice/sport drink group — The participants drink 240 mL of juice/sport drink approximately 6-8 hours after surgery
  Arms: juice/sport drink group
Dietary Supplement: Chewing gum group — The participants eat chewing gum approximately 6-8 hours after surgery
  Arms: chewing gum group

SUMMARY:
The percentage of cesarean deliveries is on the rise, accounting for 30-40% of all deliveries in Taiwan. Following a cesarean delivery, a few doctors in Taiwan still adheres to the progressive eating regimen of "nothing per mouth" for 24 hours or until the patient passes flatus or hears bowel sounds. However, a meta-analysis has shown that early oral intake (6-8 hours) significantly reduces the time required for the restoration of gastrointestinal function and hospital stay compared to delayed oral intake. Furthermore, early oral intake has not shown to increase the likelihood of gastrointestinal complications. While several food types have been adopted for early oral intake, no study has investigated the effect of different food types on clinical outcomes regarding gastrointestinal function and hospital stay for cesarean delivery. Therefore, the objective of this study is to investigate the effect of different food types on clinical outcomes for cesarean delivery through a randomized controlled trial. The subjects of this study are pregnant women who come to Chiayi Christian Hospital to schedule cesarean deliveries. They are randomly assigned to one of four groups: nothing by mouth, water, juice/sports drink, or chewing gum. The relevant clinical outcomes, such as time to first bowel sound or readiness for discharge, are recorded. One-way analysis of variance or Chi-square test is used to compare the differences among the four groups. Our expected results could provide valuable information on the type of food that could be used to improve the recovery of mothers after cesarean delivery and increase the quality of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 to 65 years
2. Receiving caesarean delivery
3. Receiving spinal and/or epidural anesthesia

Exclusion Criteria:

1. Clinical diagnosis of pre-existing gastrointestinal disorders
2. .Clinical diagnosis of an intraoperative blood loss exceeding 1000 ml during cesarean delivery
3. Clinical diagnosis of existing chronic medical disorders
4. .History of major abdominal surgery
5. Clinical diagnosis of any acute complications resulting from cesarean delivery

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
first time to bowel sound | To record the time duration from immediately after surgery to first bowel sound, an average of 24 hours.
  The investigator records the time duration of the first occurrence of bowel sounds immediately after surgery
beginning of breastmilk lactation | To record the time duration from immediately after surgery to the beginning of breast milk lactation, an average of 24 hours.
  The investigator records the time of the beginning of breast milk lactation.
length of hospital stay | To record the length of hospital stay immediately after surgery, and an average of 24 hours.
  The investigator records the length of hospital stay for each participant.

SECONDARY OUTCOMES:
time to first drink | To record the time duration from immediately after surgery to the first drink, an average of 24h.
  The investigator records the time duration of the first drink
time to first solid food intake | The time duration from immediately after surgery to the first intake of solid food, an average of 24 hours.
  The investigator measures the time it takes for the first intake of solid food.
duration of IV hydration | The time duration from immediately after surgery to IV hydration, an average of 24h.
  The investigator records the time duration of IV hydration.
IV cannulae removal | To record the time duration from immediately after surgery to IV cannulae removal, an average of 24 h.
  The investigator records the time period of IV cannulae removal.
first ambulation | To record the time duration from immediately after surgery to first ambulation, an average of 24 hours.
  The investigator records the time period of first ambulation.
first stool | To record the time period from immediately after surgery to fist stool, an average of 24 hours.
  The investigator records the time period of first stool.
satisfaction VAS (0-100) regarding the early intake | After the finish of the experiment, an average of 5 days.
  The participants report the satisfaction score (range from 0 to 100) for the early intake.

IPD SHARING:
Plan to Share IPD: No